CLINICAL TRIAL: NCT02197221
Title: IFM 2014-02 Study: A Randomized Phase III Study of Bortezomib-Melphalan 200 Conditioning Regimen Versus Melphalan 200 for Frontline Transplant Eligible Patients With Multiple Myeloma
Brief Title: Bortezomib-Melphalan Conditioning Regimen vs Melphalan for Frontline Transplant Eligible Patients With Multiple Myeloma
Acronym: IFM2014-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government); Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13 7045 01
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bortezomib-Melphalan (Experimental): Bortezomib will be administered on days: -6, -3 +1, +4. Melphalan will be administered on day -2. The PBSC will be injected on day 0.
  Interventions: Drug: Bortezomib-Melphalan
- Melphalan (Active Comparator): Melphalan will be administered on day -2. The PBSC will be injected on day 0.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Bortezomib-Melphalan — Bortezomib will be administered on days: -6, -3, +1, +4. Melphalan will be administered on day -2. The PBSC will be injected on day 0.
  Arms: Bortezomib-Melphalan
Drug: Melphalan — Melphalan will be administered on day -2. The PBSC will be injected on day 0.
  Arms: Melphalan

SUMMARY:
Phase III multicenter randomized, open-label study comparing the efficacy of a combined high dose chemotherapy using melphalan and bortezomib versus melphalan alone followed by stem cell transplant in frontline multiple myeloma patients, non-progressive after induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must have results from their initial diagnosis available at the time of screening to confirm all the following :

  1. Diagnosis of multiple myeloma according to the diagnostic
  2. Symptomatic de novo Multiple Myeloma
* Be eligible for high-dose therapy with autologous stem cell transplantation
* Autologous cell graft with a total number of CD 34 cells > or = 5 X 106/kg before freezing

Exclusion Criteria:

* Progressive disease
* Females participants pregnant or breast-feeding
* A known infection by the human immunodeficiency virus
* An active viral hepatitis B or C
* Unstable angina or myocardial infarction within 4 months prior to inclusion, heart failure NYHA class III or IV angina, uncontrolled, history of severe coronary artery disease, an uncontrolled serious ventricular arrhythmia, a sick sinus syndrome, or electrocardiographic evidence of acute ischemia or conduction disturbances grade 3 unless the patient has a pacemaker
* Uncontrolled hypertension or uncontrolled diabetes within 14 days before enrollment
* A history of another malignancy. If cancer was diagnosed more than 10 years and considered as cured, an authorization may be requested on a case-by-case basis after discussion with the principal investigator
* A significant neuropathy of grade 3-4 or grade 2 with pain in the 14 days prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Complete Response rates (according to IMWG 2011 criteria) | 60 days post Autologous Stem Cells Transplantation
overall survival | 60 months

SECONDARY OUTCOMES:
Response rates (according to IMWG 2011 criteria) | post ASCT and consolidation therapy
  Compare response rate after ASCT and after the completion of consolidation therapy
Serious adverse event | End of study
progression-free survival between the two arms | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel ATTAL, MD, PhD, Principal Investigator — University Hospital, Toulouse; Murielle ROUSSEL, MD, Principal Investigator — University Hospital, Toulouse; ROYER, MD, Principal Investigator — CHU AMIENS; DIB, MD, Principal Investigator — University Hospital, Angers; CHAOUI, MD, Principal Investigator — CH ARGENTEUIL; ARAUJO, MD, Principal Investigator — CH BAYONNE; FONTAN, MD, Principal Investigator — CH BESANCON; BRECHIGNAC, MD, Principal Investigator — HOPITAL AVICENNE BOBIGNY; MARIT, Pr, Principal Investigator — University Hospital, Bordeaux; EVEILLARD, MD, Principal Investigator — CHU BREST; MACRO, MD, Principal Investigator — CHU CAEN; MALFUSON, MD, Principal Investigator — CLAMART PERCY-Hôpital Instruction des Armées; CHALETEIX, MD, Principal Investigator — University Hospital, Clermont-Ferrand; HUMBRECHT-KRAUT, MD, Principal Investigator — Hopitaux Civils de Colmar; BELHADJ, MD, Principal Investigator — CHU Henri Mondor de Creteil; CAILLOT, MD, Principal Investigator — CHU DIJON; WETTERWALD, MD, Principal Investigator — CH DUNKERQUE; PEGOURIE, MD, Principal Investigator — University Hospital, Grenoble; AGAPE, MD, Principal Investigator — CH LA REUNION-ST DENIS; ZUNIC, MD, Principal Investigator — CH LA REUNION SAINT PIERRE; LELEU, MD, Principal Investigator — CHU LILLE; JACCARD, MD, Principal Investigator — CHU LIMOGES; KARLIN, MD, Principal Investigator — Hospices Civils de Lyon; NICOLAS, MD, Principal Investigator — Centre Léon Bérard de LYON; STOPPA, MD, Principal Investigator — Institut Paoli Calmettes, Marseille; DORVAUX, MD, Principal Investigator — CH METZ; EISENMANN, MD, Principal Investigator — CH Mulhouse; HULIN, MD, Principal Investigator — CHU NANCY; MOREAU, Pr, Principal Investigator — Nantes University Hospital; LEGROS, MD, Principal Investigator — CHU NICE; BENBRAHIM, MD, Principal Investigator — CH ORLEANS; BOUSCARY, MD, Principal Investigator — Hôpital Cochin Paris; KUHNOWSKI, MD, Principal Investigator — Institut Curie Paris; MOREL, MD, Principal Investigator — Hôpital la Pitié Salpêtrière Paris; GARDERET, MD, Principal Investigator — Hôpital Saint Antoine Paris; ARNULF, MD, Principal Investigator — Hôpital Saint Louis Paris; LACOTTE, MD, Principal Investigator — CHU Poitiers; DELMER, Pr, Principal Investigator — CHU REIMS; ESCOFFRE, MD, Principal Investigator — CHU Rennes; LENAIN, MD, Principal Investigator — Centre Henri Becquerel de Rouen; GLAISNER, MD, Principal Investigator — Hôpital René Huguenin - St Cloud; AUGEL MEUNIER, MD, Principal Investigator — CHU ST PRIEST EN JAREZ; BENBOUBKER, MD, Principal Investigator — CHU Tours; RIGAUDEAU, MD, Principal Investigator — CH Versailles
Locations (46):
- Belgium (4):
  - Clinique Universitaire Saint Luc, Brussels
  - Grand Hôpital de Charleroi - Site Notre-Dame, Charleroi
  - Chu Liege, Liège
  - CHU Dinant-Godinne UCL Namur, Yvoir
- France (42):
  - Hôpital Felix Guyon, Saint-Denis, ILE de LA Reunion
  - CH sud Réunion, Saint-Pierre, ILE de LA Reunion
  - CHU Amiens, Amiens
  - Chu Angers, Angers
  - CH Argenteuil Victor Dupouy, Argenteuil
  - CH Bayonne, Bayonne
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Avicenne, Bobigny
  - Hôpital du Haut Lévêque, Bordeaux
  - CHU DE BREST Hôpital A.Morvan, Brest
  - CHU CAEN, Caen
  - Hôpital d'instruction des armées Percy, Clamart
  - CHU d'Estaing, Clermont-Ferrand
  - Hôpitaux civils de Colmar, Colmar
  - CHU Henri Mondor, Créteil
  - CHRU Dijon - Hôpital des Enfants, Dijon
  - Centre Hospitalier Général, Dunkirk
  - CHU Grenoble, Grenoble
  - CHRU LILLE- Hôpital Claude Huriez, Lille
  - Chu Limoges, Limoges
  - Centre Hospitalier Lyon sud, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital de Mercy - CHR Metz Thionville, Metz
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Chu Nancy, Nancy
  - Hôtel Dieu, Nantes
  - Hôpital Archet, Nice
  - CH d'Orléans, Orléans
  - Hôpital Cochin, Paris
  - Hôpital de la Pitié Salpêtrière, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital St-Antoine, Paris
  - CHU - Hôpital Jean Bernard, Poitiers
  - CHU de Reims- Hôpital R.Debré, Reims
  - Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Hôpital René Huguenin, Saint-Cloud
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - CHU de Toulouse, Toulouse
  - Chu Tours, Tours
  - Centre Hospitalier de Versailles-Hôpital André Mignot, Versailles

REFERENCES:
- [Result] Roussel M, Lauwers-Cances V, Macro M, Leleu X, Royer B, Hulin C, Karlin L, Perrot A, Touzeau C, Chretien ML, Rigaudeau S, Dib M, Nicolas-Virelizier E, Escoffre-Barbe M, Belhadj K, Mariette C, Stoppa AM, Araujo C, Doyen C, Fontan J, Kolb B, Garderet L, Brechignac S, Malfuson JV, Jaccard A, Lenain P, Borel C, Hebraud B, Benbrahim O, Dorvaux V, Manier S, Augeul-Meunier K, Vekemans MC, Randriamalala E, Chaoui D, Caers J, Chaleteix C, Benboubker L, Vincent L, Glaisner S, Zunic P, Slama B, Eveillard JR, Humbrecht-Kraut C, Morel V, Mineur P, Eisenmann JC, Demarquette H, Richez V, Vignon M, Caillot D, Facon T, Moreau P, Colin AL, Olivier P, Wuilleme S, Avet-Loiseau H, Corre J, Attal M. Bortezomib and high-dose melphalan conditioning regimen in frontline multiple myeloma: an IFM randomized phase 3 study. Blood. 2022 May 5;139(18):2747-2757. doi: 10.1182/blood.2021014635. PMID 35511184